CLINICAL TRIAL: NCT06465433
Title: An Open-Label, Multicenter, Extension Study to Provide Continued Treatment for Patients With Hematologic Malignancies Previously Enrolled in Studies With Tafasitamab
Brief Title: Extension Study to Provide Continued Treatment for Patients With Hematologic Malignancies Previously Enrolled in Studies With Tafasitamab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR208C216; 2022-500765-27-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — tafasitamab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tafasitamab Dose (Experimental): Treatment with tafasitamab is as per the treatment dose and schedule they received in the parent protocols.
  Interventions: Drug: Tafasitamab

INTERVENTIONS:
Drug: Tafasitamab — Treatment with tafasitamab is as per the treatment dose and schedule they received in the parent protocols.

SUMMARY:
This extension study is designed to enroll participants with hematologic malignancies who are receiving clinical benefit from tafasitamab treatment in a parent study with tafasitamab..

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Having been enrolled and is still receiving treatment with tafasitamab at the end of a parent tafasitamab clinical study.
* Is tolerating tafasitamab treatment at the dose specified in the parent protocol as assessed by the Investigator.
* Is in complete/partial response or stable disease and is receiving clinical benefit from treatment with tafasitamab in the parent study, as assessed by the Investigator.
* Has demonstrated compliance, as assessed by the Investigator, with the parent protocol requirements.
* Willingness and ability to comply with scheduled visits, treatment plans, and any other study procedures indicated in this protocol.

Exclusion Criteria:

* Patient who is legally institutionalized, or under judicial protection.
* Has met one or more criteria for permanent tafasitamab treatment discontinuation as stipulated in the parent protocol.
* Able to access tafasitamab outside a clinical study.
* Patient with an uncontrolled intercurrent illness or any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.
* A female patient who is pregnant confirmed by a pregnancy test prior to enrollment, breastfeeding, or a woman of childbearing potential (WOCBP) who does not agree to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of study treatment, and does not refrain from donating oocytes during this period.
* A male patient who does not agree to use contraception as detailed in the contraceptive guidance during the treatment period and for at least 3 months after the last dose of study treatment (if they have a heterosexual partner who is a woman of childbearing potential) and who does not refrain from donating sperm during this period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-08-29 (Estimated); Study Completion 2027-08-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | up to approximately 2 years
  Defined as any Adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug up to 90 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Director, Study Director — Incyte Corporation
Locations (5):
- Petz Aladar County Teaching Hospital, Győr, Hungary
- Hospital S.M. Terni University of Perugia, Terni, Italy
- Samsung Medical Center, Seoul, South Korea
- Clinica Universitad de Navarra, Pamplona, Spain
- Gazi University Hospital Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Extension Study to Provide Continued Treatment for Patients With Hematologic Malignancies Previously Enrolled in Studies With Tafasitamab — https://incyteclinicaltrials.com/studies/mor208c216